CLINICAL TRIAL: NCT02716740
Title: Pilot Study of Branched Amino Acid Supplementation for Patients With an Excessive Loss of Muscular Body Mass After Obesity Surgery.
Brief Title: Study of Amino Acid Supplementation for Patients With an Excessive Loss of Muscular Body Mass After Obesity Surgery.
Acronym: MUSCAADE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patient
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RC31/15/7649; 2015-A01226-43 (Other: RCB)
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Post-obesity surgery; Leucine-enriched amino acid supplementation; Anabolic substance; Physical training; Muscular mass; Loss of weight
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucine-enriched amino acid : 2.16g/day (Experimental): Dietary Supplement: Leucine-enriched amino acid supplementation and 30 minutes of physical training 3 times per week (2.16g/day)
  Interventions: Dietary Supplement: Leucine-enriched amino acid supplementation and 30 minutes of physical training 3 times per week
- Leucine-enriched amino acid : 4g/day (Experimental): Dietary Supplement: Leucine-enriched amino acid supplementation and 30 minutes of physical training 3 times per week (4g/day).
  Interventions: Dietary Supplement: Leucine-enriched amino acid supplementation and 30 minutes of physical training 3 times per week

INTERVENTIONS:
Dietary Supplement: Leucine-enriched amino acid supplementation and 30 minutes of physical training 3 times per week — After 3 months of obesity-surgery, if patients lost more than 15% of muscular weight, they will take a leucine-enriched amino acid supplementation during 3 months added with a regular physical training (30 minutes, 3 times/week). Arm A will take 2.46g/day of leucine-enriched amino acid supplementation and arm B 4g/day.

SUMMARY:
Despite the demonstrable health and quality of life benefits, there are unknowns within consequences of obesity surgery. Weight loss composition is poorly understood. The objective is to have a significant loss of body fat and a limited loss of muscular weight.

A cohort study in the nutrition unit at Toulouse University Hospital shows that 3 months and 1 year after surgery, there are 2 phenotypes of patients. The first one is called 'little loss' and is defined by a contribution of muscular weight lower than 15% of the total weight loss. The other one is called 'big loss' and is defined by a contribution of muscular weight higher than 15% of the total weight loss. Causes of these different phenotypes are unknown for the moment.

Some amino acids have an anabolic potential. Leucine induces a muscular protein synthesis in clinical situations like hepatic cirrhosis, and some populations like new born and older people.

Assuming that, a leucine-enriched essential amino acid supplementation will have a benefit effect on the muscular mass. That is testing the influence of the quality of protein consumed, more than the quantity. An anabolic substance (amino acid here) can lead to gain of muscle only if it is associated to regular physical training, all patients will follow a physical training.

DETAILED DESCRIPTION:
An excessive loss of lean mass could have negative metabolic consequences. Indeed, lean mass is an essential determinant of weight loss and of the glycaemia regulation. An important loss of muscular mass could expose the person to a reduction of quality of life (because of fatigue), or even a functional loss. Muscles are important for insulin sensibility and glucose metabolism. Muscles are proteolysis target and proteins will be used as sources of amino acid for other cellular functions.

Changes in lean mass have been at the centre of several studies, but changes in muscular mass after bariatric surgery have been report only one time.

A cohort study in the nutrition unit at Toulouse University Hospital shows that 3 months and 1 year after surgery, there are 2 phenotypes of patients. The first one is called 'little loss' and is defined by a contribution of muscular weight lower than 15% of the total weight loss. The other one is called 'big loss' and is defined by a contribution of muscular weight higher than 15% of the total weight loss. Causes of these different phenotypes are unknown for the moment. Nothing distinguishes them before the surgery. Type of surgery, gender, protein intake (in grams of proteins intake per day) do not appear to have a determining influence about the intensity of muscle mass loss. The only other study published shows changes in muscular mass about 15% at 6 weeks.

Relation between glycaemia changes and muscle mass changes suggests that patients with modest changes in muscular mass are patients who have the best improvement of glycaemia after surgery. It is the reason why, it could be interesting to preserve muscular mass.

Nowadays, there is no consensual strategy to compensate this loss of muscle mass. It is important to have in the same time an anabolic stimulus (training, hormone…) and a sufficient energy and protein intake.

According to a recent study which compares leucine intake with placebo during weight loss driven by a low-calorie diet associated to a muscle strengthening exercises, patients loss the same weight, but leucin group is gaining lean mass, while placebo group is losing it. Accordingly, twe different doses of amino acid will be tested of those used as diet supplement.

This study is testing the influence of the quality of protein consumed, more than the quantity. Patients will take leucine-enriched amino acid supplement and follow physical training. Aromatic amino acid supplementation showed an anabolic effect in older people, undernourished children and undernourished patients with chronic obstructive pulmonary disease. There are no known side effects. This amino acid supplementation has not been evaluated in post-obesity surgery context.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years of age and younger than 65 years of age,
* Patient received an obesity-surgery (gastric bypass or sleeve gastrectomy)
* Contribution of muscular weight higher than 15% of the total weight loss after the third month post-surgery.
* Patient that be able to increase their physical activity
* Patient that give their informed consent before any procedure for the study
* Patient affiliated with a health insurance scheme

Exclusion Criteria:

* Patients allergic to one of the supplement's compound.
* Patients with glucocorticoid therapy
* Patients with hyperthyroidism
* Patients commencing insulin treatment or growth hormone
* Protein powder intake (as nutritional complement or as anabolic substance for muscle building practice)
* Oral nutritional supplement intake for malnutrition
* Bone fracture since the surgery
* Infection can cause hypercatabolism (like microbial outbreak or chronic gastric fistula)
* Hospitalization for more than 24 hours since the surgery
* Known physical handicap
* Inability to increase physical activity during 3 months after beginning of the supplementation
* Enteral or parenteral nutrition
* Patients over 158 kg (DEXA impossible)
* Protected adults (guardianship by court order)
* Pregnant woman or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in appendicular muscular mass at 3 months | Baseline and 3 months
  Appendicular muscular mass measured by dual-energy X-ray absorptiometry (DEXA). It will be measured before and 3 months after supplementation.

SECONDARY OUTCOMES:
Change from baseline in limbs muscular force at 3 months | Baseline and 3 months
  The lower and higher limbs muscular force will be measured with a strain gauge.
Change from baseline in muscular function at 3 months | Baseline and 3 months
  400 meters walking speed
Change from baseline in muscular function at 3 months | Baseline and 3 months
  Chair-stand test
Change from baseline in muscular function at 3 months | Baseline and 3 months
  Balance test by the Short Physical Performance Battery test
Change from baseline in fatigue at 3 months | Baseline and 3 months
  Fatigue will be evaluate by the Pichot scale
Change from baseline in general functional assessment at 3 months | Baseline and 3 months
  General function will be assessed by the Functional Status Questionnaire test.
Change from baseline in protein daily intake at 3 months | Baseline and 3 months
  Patient will evaluate his/her protein daily intake (in g/day) by the Protein Intake Monitor with a digital tablet
Change from baseline in physical training adhesion at 3 months | Baseline and 3 months
  Patients will have an exercise diary to write their organised physical activity. Physical activity will be converted in a multiple of basal metabolic rate.
Change from baseline in glucose metabolism at 3 months | Baseline and 3 months
  Oral glucose tolerance test will be performed and glucose concentration will be determined into the blood.
Change from baseline in insulin secretion at 3 months | Baseline and 3 months
  Oral glucose tolerance test will be performed and insulin concentration will be determined into the blood.
Change from baseline in leucine compliance | Baseline and 3 months
  Leucine concentration and variation between visit before and after 3 months of supplementation will be measured by chromatography to assess the patient's compliance

CONTACTS AND LOCATIONS:
Overall Officials: RITZ Patrick, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Department of Endocrinology, metabolic diseases and nutrition, Toulouse, France

IPD SHARING:
Plan to Share IPD: No